CLINICAL TRIAL: NCT06290999
Title: Study of Multifrequential Impedancemetry in Pulsatile Tinnitus
Acronym: MADMAN
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2023/80
Record Dates: First submitted 2024-02-26; First posted 2024-03-04 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Pulsatile Tinnitus
Keywords: Pulsatile Tinnitus; multifrequency admittancemetry
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patient with pulsatile tinnitus
  Interventions: Diagnostic Test: multifrequential admittancemetry

INTERVENTIONS:
Diagnostic Test: multifrequential admittancemetry — Every participant of the study have to complete an Ear, Nose and Throat examination included a conventional audiometry, and a multifrequential admittancemetry.
  if radio-interventional venous stenting is not indicated, an multifrequential admittancemetry will also be performed 3 months after the procedure.

SUMMARY:
This study intended to search for a relationship between the multifrequential admittancemetry and the pulsatile tinnitus.

DETAILED DESCRIPTION:
The multifrequency admittancemetry is known to reflect several parameters of the middle ear and the external ear. More recently it appears to also reflect some parameters of the inner ear, such as the perilymph pressure. Furthermore, investigators do not know exactly the physiopathology of pulsatile tinnitus that are from veinous etiology. Modifications of the perilymphatic pressure could be implicated. Investigators intended to search for a relationship between these both theories.

Investigators will include every patient that consult to Ear, Nose and Throat unit of Bordeaux University Hospital with a pulsatile tinnitus trouble, and perform multifrequential admittancemetry. If a radio-surgical intervention is scheduled for a venous stenosis, the test will also be performed test after the surgery.

If there is no surgical intervention, no follow-up will be required.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient
* Unilateral or bilateral pulsatile tinnitus
* Pulsatile tinnitus > 1 month old
* Affiliated or beneficiary of by social security system

Exclusion Criteria:

* Otological surgery, excluding trans-tympanic aerators in childhood with closed eardrum
* Middle ear abnormality (any type of partial or total filling of the middle ear) noted on otoscopy or subsequent MRI scan
* Abnormal eardrums excluding tympanosclerosis
* Non-pulsatile tinnitus
* Conductive hearing loss with abolition of stapedial reflexes
* Minor patient
* Major protected
* Abnormal tympanometry at 226 Hz
* Presence of rotatory vertigo
* Opposition to participation expressed by patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Unilateral or bilateral pulsatile tinnitus
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-06-03 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Multifrequency admittancemetry | At Day 0 (inclusion)
  G conductance peak width at 2000 Hz

SECONDARY OUTCOMES:
compression maneuvers | At Day 0 (inclusion)
  Evaluation of the effect of compression maneuvers on the width of the G 2000 peak of the IMF in venous or arterial pulsatile tinnitus, whether or not the maneuver is effective.
Evaluation of the effect of interventional radiology | up to 3 month after inclusion (M3)
  Evaluation of the effect of interventional radiology procedures such as transverse sinus stenting on MFI values.
success of radiointerventional treatment | up to 3 month after inclusion (M3)
  Search for a predictive factor of success of radiointerventional treatment of venous pulsatile tinnitus: search for a threshold value of pre-operative G2000, separating two groups: success and non-success (groups defined by a THI (Tinnitus Handicap Index) divided by 2 in the success group).

CONTACTS AND LOCATIONS:
Locations (1):
- Bordeaux University Hospital, Bordeaux, France